CLINICAL TRIAL: NCT03742375
Title: Quantitative HPV Genotyping in Screening of Anal Intraepithelial Neoplasia in HIV-positive Patients
Acronym: GAIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Sciensano (Other Government)
Responsible Party: Principal Investigator, prof. dr. Philip Roelandt, Assistant head of clinic Gastroenterology, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S60050
Record Dates: First submitted 2018-10-10; First posted 2018-11-15 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Human Immunodeficiency Virus
Keywords: Human Papilloma Virus; Anal Intraepithelial Neoplasia
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV genotyping (Experimental)
  Interventions: Diagnostic Test: HPV genotyping

INTERVENTIONS:
Diagnostic Test: HPV genotyping — Quantitative HPV genotyping on anal swab

SUMMARY:
The pathophysiology from anal HPV infection to Anal Intraepithelial Neoplasia is less well understood than cervical HPV infection. In cervical screening programs it is well accepted that the sole presence of a high-risk HPV strain (irrespective of number of viral particles) is sufficient to justify further investigation and treatment. The investigators hypothesize that in anal HPV infection not only the presence but the extent of HPV infection (single genotype viral load) or combination of different HPV genotypes (cumulative viral load) is of importance in determining the risk of anal dysplasia.

ELIGIBILITY:
Inclusion criteria

* Stable HIV disease (i.e. receiving ART for at least 1 year, no adverse drug reactions requiring regular monitoring, no current illnesses or pregnancy, good understanding of lifelong adherence and evidence of treatment success: two consecutive undetectable viral load measures)
* Referred for high-resolution anoscopy

Exclusion criteria

* Documented AIN (treated or untreated)
* Local anal inflammation (proctitis) and/or acute fissure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of HPV subtypes in HIV-positive patients | 1 minute
  Retrieval of 1 anal swab before performing HRA to determine the HPV subtypes at that particular moment

SECONDARY OUTCOMES:
Correlation between high-resolution anoscopy findings and quantitative HPV genotyping | 30 minutes up to 10 days
  Performing HRA (30 minutes) with or without biopsies, results biopsies up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Philip Roelandt, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No